CLINICAL TRIAL: NCT00634296
Title: The Effects of the Inspiratory Muscle Training Plus Aerobic Training Compare to Aerobic Training Alone in Heart Failure Patients With Inspiratory Muscle Weakness.
Brief Title: The Effects of the Inspiratory Muscle Plus Aerobic Training Compare to Aerobic Training Alone in Heart Failure Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Jorge Pinto Ribeiro, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCPA2004-302
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Heart Failure
Keywords: Heart failure; Systolic dysfunction; Inspiratory muscle weakness
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G2 (Active Comparator): Inspiratory muscle training added by aerobic training to aerobic training alone
  Interventions: Other: Inspiratory muscle added by aerobic to aerobic alone

INTERVENTIONS:
Other: Inspiratory muscle added by aerobic to aerobic alone — Inspiratory muscle added by aerobic to aerobic alone
  Other Names: Aerobic: G1; Inspiratory muscle added by aerobic: G2

SUMMARY:
This study aims to compare effects of inspiratory muscle training added by aerobic training to aerobic training alone in heart failure patients with inspiratory muscle weakness. To do so, strength and endurance of inspiratory muscles, functional capacity, quality of life, heart rate variability and sleep apnea evaluations will be conducted in patients with heart failure.

DETAILED DESCRIPTION:
A sample comprising at least 30 individuals is necessary. These subjects will be randomized in two groups, one consisting of inspiratory muscle training plus aerobic training, whereas the other will consist of the aerobic training alone.

This prospective, randomized, controlled trial will include patients with the diagnosis of chronic heart failure attributable to left ventricular systolic dysfunction who will be recruited from the Heart Failure Clinic.

Entry criteria for the study are a previous history of symptomatic heart failure caused by left ventricular systolic dysfunction, inspiratory muscle weakness (PImax < 70% of the predicted), and clinical stability, including no change in medications for the past three months.

Exclusion criteria will be unstable angina, myocardial infarction, or cardiac surgery within the previous three months, chronic metabolic, orthopedic, or infectious diseases, treatments with steroids, hormones, or cancer chemotherapy, history of exercise-induced asthma, chronic obstructive pulmonary disease and smokers will be not recruited.

The protocol was approved by the Committee for Ethics in Research of Hospital de Clinics de Porto Alegre and Ijuí University and all subjects are required to sign an informed consent form.

Variables will be measured by strength and endurance (progressive and constant load), 6-min walk test, cardiopulmonary exercise testing, quality of life questionnaire, evaluation of the heart rate variability and sleep apnea.

The inspiratory muscle training plus aerobic training will consist of cycle exercise (3 sessions/week) and inspiratory exercise by using Threshold equipment for 30 min, 7 times per week, whereas aerobic training group will perform only cycle exercise. Both treatments will last 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* previous history of symptomatic heart failure caused by left ventricular systolic dysfunction
* inspiratory muscle weakness (PImax < 70% of the predicted)
* clinical stability, including no change in medications for the past three months

Exclusion Criteria:

* unstable angina
* myocardial infarction, or cardiac surgery within the previous three months
* chronic metabolic, orthopedic, or infectious diseases
* treatments with steroids, hormones, or cancer chemotherapy
* history of exercise-induced asthma, chronic obstructive pulmonary disease
* smokers

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-03; Primary Completion 2008-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To compare effects of inspiratory muscle training added by aerobic training to aerobic training alone in heart failure patients with inspiratory muscle weakness. | one year

SECONDARY OUTCOMES:
To compare effects between the training groups evaluating strength and endurance of inspiratory muscles; functional capacity; the physical and psychological perceptions of quality of life and heart rate variability and sleep apnea. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jorge P. Ribeiro, MD, ScD, Principal Investigator — Associate Professor and Chief of Non-invasive Cardiology
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Winkelmann ER, Chiappa GR, Lima CO, Viecili PR, Stein R, Ribeiro JP. Addition of inspiratory muscle training to aerobic training improves cardiorespiratory responses to exercise in patients with heart failure and inspiratory muscle weakness. Am Heart J. 2009 Nov;158(5):768.e1-7. doi: 10.1016/j.ahj.2009.09.005. Epub 2009 Oct 2. PMID 19853695